CLINICAL TRIAL: NCT02036229
Title: a Randomised, Double Blind, Placebo Controlled, Half- Face Study to Evaluate the Effect of Topical Ivermectin Cream 0.5% on Demodicidosis
Brief Title: Topical 0.5% Ivermectin Cream for Treatment of Demodicidosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Rina Segal, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: topical ivermectin, demodex
Record Dates: First submitted 2014-01-02; First posted 2014-01-14 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Demodicidosis; Rosacea
Keywords: demodex; demodicidosis; rosacea; ivermectin
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5% ivermectin cream (Experimental): Each participant will be treated with topical ivermectin cream 0.5% qd for one half of the face for 1 month. In the second month all patients will be treated with ivermectin cream for the entire skin involvement.
  Interventions: Drug: ivermectin cream 0.5%
- vehicle cream (Placebo Comparator): Each participant will be treated with a vehicle cream qd for the other half of the face for 1 month. In the second month all patients will be treated with ivermectin cream for the entire skin involvement.
  Interventions: Drug: ivermectin cream 0.5%

INTERVENTIONS:
Drug: ivermectin cream 0.5% — Each participant will be treated with topical ivermectin cream 0.5% qd for one half of the face and with a vehicle cream qd for the other half of the face for 1 month. In the second month all patients will be treated with ivermectin cream for the entire skin involvement.

SUMMARY:
The purpose of this study is to determine whether 0.5% ivermectin cream is effective in the treatment of demodicidosis (including papulopustular rosacea)

ELIGIBILITY:
Inclusion Criteria:

* subjects with clinical and laboratory diagnosis of demodicidosis with symmetrical facial eruption who are willing to comply with study requirements

Exclusion Criteria:

* known hypersensitivity to ivermectin.
* pregnancy
* immunodeficiency such as HIV or immunosuppressive therapy
* concomitant use of systemic antibiotics or steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
A decrease in mite density in skin surface biopsy after treatment with topical ivermectin (≤5 mites/cm2 for skin lesions). | 5 months

SECONDARY OUTCOMES:
Clinical improvement | 5 months
  Clinical improvement will be assessed by objective evaluation of erythema, dryness, scaling, roughness, and/or papules/pustules in skin lesions and subjective evaluation of itch and dryness.
A comparable dermoscopic improvement in the demodicidosis features | 5 months
  dermoscopic demodicidosis features:
  * number of demodex tails
  * demodex follicular openings
  * reticular dilated vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Segal, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- RabinMC, Dermatology dept., Petah Tikva, Israel